CLINICAL TRIAL: NCT06078306
Title: Clinical Trial for the Safety and Efficacy of Induction Chemotherapy With Azacitidine+Venetoclax (VA) and Bridging CD19CD22 CAR-T Therapy in Adult Patients With Newly Diagnosed High-Risk and Ph-negative (Ph-) B-ALL
Brief Title: CD19CD22 CAR-T Therapy in Patients With High-Risk B Acute Lymphoblastic Leukemia (B-ALL).
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: High Risk B-ALL
Record Dates: First submitted 2023-09-11; First posted 2023-10-11 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2023-10

CONDITIONS: B Acute Lymphoblastic Leukemia; Ph-Negative ALL; High Risk Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Burkitt Lymphoma | interventions — Azacitidine; venetoclax

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR-T therapy (Experimental): Therapeutic outcomes in adults with Ph- B-ALL have substantially improved in the last decade, with complete remission (CR) and long-term overall survival (OS) rates of around 90% and 40%-50%, respectively. The presence of measurable residual disease (MRD) is the strongest predictor of relapse in B-ALL. In this study, high risk Ph- B-ALL patients receive the induction chemotherapy with Azacitidine+Venetoclax. After induction chemotherapy with Azacitidine+Venetoclax (VA regime), each subject receives CD19CD22 CAR-T cells by intravenous infusion. The patients with MRD negative will undergo HSCT.
  Interventions: Drug: Azacitidine Injection; Drug: Venetoclax; Drug: CD19CD22 CAR-T

INTERVENTIONS:
Drug: Azacitidine Injection — Azacitidine Injection 75mg/square meter/day, day1-7, subcutaneous injection
  Other Names: Azacitidine
Drug: Venetoclax — Venetoclax 100mg day 1, 200mg day 2, 400mg d3-d21, oral
  Other Names: ABT-199
Drug: CD19CD22 CAR-T — After induction chemotherapy with Azacitidine+Venetoclax, each subject receives CD19CD22 CAR-T cells by intravenous infusion
  Other Names: GDC-0199

SUMMARY:
Clinical trial for the safety and efficacy of induction chemotherapy with VA regime and bridging CD19CD22 CAR-T therapy in adult patients with newly diagnosed high-risk and Ph- B-ALL

DETAILED DESCRIPTION:
To evaluate the safety and efficacy of induction chemotherapy with VA regime and bridging CD19CD22 CAR-T therapy in Adult patients with newly diagnosed high-risk and Ph- B-ALL in this prospective, single arm study.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18 and ≤65 years old
2. Newly diagnosed and high risk B-ALL according to the 2022 WHO classification
3. The immunophenotype of leukemia cells were CD19 and CD22 positive and Ph-;
4. Anticipated survival time more than 12 weeks;
5. Those who voluntarily participated in this trial and provided informed consent.

Exclusion Criteria:

1. History of craniocerebral trauma, conscious disturbance, epilepsy, cerebrovascular ischemia, and cerebrovascular hemorrhagic diseases;
2. Electrocardiogram shows prolonged QT interval, severe heart diseases such as severe arrhythmia in the past;
3. Pregnant (or lactating) women;
4. Patients with severe active infections (excluding simple urinary tract infection and bacterial pharyngitis);
5. Human immunodeficiency virus (HIV) positive; Active infection of hepatitis B virus or hepatitis C virus
6. Previously treated with any CAR-T cell product or other genetically-modified T cell therapies;
7. Creatinine>2.5mg/dl, or ALT / AST > 3 times of normal amounts, or bilirubin>2.0 mg/dl;
8. Other uncontrolled diseases that were not suitable for this trial;
9. Any situations that the investigator believes may increase the risk of patients or interfere with the results of study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-04-20 (Estimated); Primary Completion 2024-09-10 (Estimated); Study Completion 2025-09-10 (Estimated)

PRIMARY OUTCOMES:
Complete Remission Rate | The cycle of CD19CD22 cell therapy is day 2-4; Effect evaluation was day 21 after CD19CD22 cells infusion
  MRD Negative Remission Rate after CD19CD22 cell therapy

SECONDARY OUTCOMES:
Complete Remission Rate of VA regime | The cycle of VA regime is day 21; Effect evaluation was day 7 after VA regime
  Complete Remission Rate after VA regime
Complete Molecular Remission Rate | The cycle of CD19CD22 cell therapy is day 2-4; Effect evaluation was day 21 after CD19CD22 cells infusion
  Complete Molecular Remission Rate after CD19CD22 CAR-T cell therapy
Overall survival (OS) | The cycle of CD19CD22 cell therapy is day 2-4; Effect evaluation was 2 years after CD19CD22 CAR-T cells infusion
  From the first infusion of CD19CD22 cells to death or the last visit
Leukemia-free survival (LFS) | The cycle of CD19CD22 cell therapy is day 2-4; Effect evaluation was 2 years after CD19CD22 CAR-T cells infusion
  Up to 2 years after CD19CD22 CAR-T cells infusion

CONTACTS AND LOCATIONS:
Locations (1):
- Xiaowen Tang, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No